CLINICAL TRIAL: NCT03058016
Title: Personalized Nutrition Prediction for Metabolic Syndrome Patients, an Open Single-center Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Galilee CBR (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 98-16
Record Dates: First submitted 2017-02-07; First posted 2017-02-20 (Actual); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Diet

STUDY DESIGN:
Intervention Model Description: Personalized recommendations for effective diet, lifestyle and activities based on the patient's parameters measurements and reactions will be provided on a bi-weekly basis, all Lab tests and dietician control will be performed twice a month.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Personalized recommendations for diet (Experimental): After measurement of individual's parameters changes as blood tests, gut microbiome, urine tests, blood pressure, heart performance, body circumferences, mood and mental status as well as monitoring each individual's food intake - a model to predict individual's body reaction according to lifestyle, eating and activity habits will be built.
  Personalized recommendations for effective diet, lifestyle and activities based on the patient's parameters measurements and reactions will be provided on a bi-weekly basis, all Lab tests and dietician control will be performed twice a month.
  Interventions: Other: Personalized recommendations for diet

INTERVENTIONS:
Other: Personalized recommendations for diet — Personalized recommendations for effective diet, lifestyle and activities based on the patient's parameters measurements and reactions

SUMMARY:
This clinical study is designed to evaluate the providing of a computational prediction engine for optimization of personalized nutrition

Personalized recommendations for effective diet, lifestyle and activities based on the patient's parameters measurements and reactions will be provided on a bi-weekly basis, all Lab tests and dietician control will be performed twice a month.

DETAILED DESCRIPTION:
Pre-diabetic and pre-metabolic syndrome patients will be recruited to the study for a period of one year.

After measurement of individual's parameters changes as blood tests, gut microbiome, urine tests, blood pressure, heart performance, body circumferences, mood and mental status as well as monitoring each individual's food intake - a model to predict individual's body reaction according to lifestyle, eating and activity habits will be built.

Personalized recommendations for effective diet, lifestyle and activities based on the patient's parameters measurements and reactions will be provided on a bi-weekly basis, all Lab tests and dietician control will be performed twice a month.

ELIGIBILITY:
Inclusion Criteria:

1. Adults age 18-65
2. HBA1C between 5.5 and 7%.
3. Altered lipid metabolism
4. BMI > 25
5. Signed Informed Consent

Exclusion Criteria:

1. Pregnancy
2. Usage of antibiotics within three months prior to participation
3. Chronically active inflammatory or neoplastic disease in the three years prior to enrollment
4. Chronic gastrointestinal disorder, including Inflammatory Bowel Disease and Celiac Disease
5. Skin disease, including contact dermatitis, precluding proper attachment of the continuous glucose monitor
6. Active psychiatric disorder
7. Myocardial infarction or cerebrovascular accident in the 6 months prior to participation
8. Chronic immunosuppressive medication usage
9. Clinical depression

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2017-04-01 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
To determine number of participants with reduced BMI | One year
  Change at 12 months
To determine number of participants with reduced hA1C | One year
  Change at 12 months
To determine number of participants with reduced cholesterol | One year
  Change at 12 months

SECONDARY OUTCOMES:
Type of intestinal microorganisms | One year
  The participants microbiome will be analyzed before and after the trial. The type of microorganisms will be determined by microbiological measurements.
Number of intestinal microorganisms | One year
  The participants microbiome will be analyzed before and after the trial. The number of microorganisms will be determined by microbiological measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Keren, Study Director — 972545413328

IPD SHARING:
Plan to Share IPD: No